CLINICAL TRIAL: NCT01415219
Title: Efficacy of an Individual Rehabilitation Program in Polymyositis and Dermatomyositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007_0712; 2007-A00756-47 (Other: ID-RCB number, AFSSAPS); PHRC 2006/1916 (Other: DHOS); DGS 2007-0440 (Other: AFSSAPS)
Record Dates: First submitted 2010-04-08; First posted 2011-08-11 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2014-12

CONDITIONS: Dermatomyositis; Polymyositis
Keywords: rehabilitation; exercise; efficacy; functional status
MeSH Terms: conditions — Dermatomyositis; Polymyositis; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active rehabilitation (Active Comparator): A program of 12 individual exercise sessions (3 per week during 4 weeks)
  Interventions: Other: Active rehabilitation
- conventional care (No Intervention): community based physiotherapy

INTERVENTIONS:
Other: Active rehabilitation — A program of 12 individual exercise sessions (3 per week during 4 weeks)
  Arms: active rehabilitation

SUMMARY:
The purpose of this study is to evaluate the efficacy of an active rehabilitation program on disability and quality of life of patients affected by dermatomyositis and polymyositis.

DETAILED DESCRIPTION:
Dermatomyositis (DM) and polymyositis (PM) are inflammatory disabling neuromuscular disorders. Despite partial benefit of pharmacological treatments, muscle strength, functional status and quality of life remain impaired. Although the use muscle exercises in (DM) and (PM) have been reported, its efficacy on disability and quality of life has not been proved.

Te aim of the study is to evaluate the benefit at mid term (12 months) of an active rehabilitation program administrated to patients affected by PM and DM.

Method: a 3 year prospective, multicentric, randomized controlled trial A program of 12 individual exercise sessions (3 per week during 4 weeks) is compared to conventional care. Patients are followed 12 month after the inclusion.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Dermatomyositis ore polymyositis according to the International Myositis Assessment and Clinical Studies Group
* functional impairment (an HAQ score greater than 0.5)
* stability of muscle impairment
* medical insurance

Exclusion Criteria:

* no recent inflammatory activity
* other chronic disease
* cognitive impairment
* patients who participated to a rehabilitation program before inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-03; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
HAQ score | 6 month and 1 year after rehabilitation

SECONDARY OUTCOMES:
Quality of life (SF36 score) | 6 month and 1 year after rehabilitation
MFM(motor function measure) | 6 month and one year after rehabilitation
muscle strength (MRC manual muscle testing) | at 6 month and one year after rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Andre Thevenon, Professor, Principal Investigator — University Hospital, Lille
Locations (5):
- France (5):
  - University Hospital, Lille, Lille, Hauts-de-France
  - Hopital Rotschild, Paris
  - GH Pitié Salpétrière, Paris
  - Hopital Cochin, Paris
  - Centre hospitalier universitaire de Rouen, Rouen

REFERENCES:
- [Result] Tiffreau V, Rannou F, Kopciuch F, Hachulla E, Mouthon L, Thoumie P, Sibilia J, Drumez E, Thevenon A. Postrehabilitation Functional Improvements in Patients With Inflammatory Myopathies: The Results of a Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Feb;98(2):227-234. doi: 10.1016/j.apmr.2016.09.125. Epub 2016 Oct 24. PMID 27789240